CLINICAL TRIAL: NCT02448433
Title: Phototherapy in Young People With Depression; Investigating Associations Between Changes in Actigraphic Sleep-wake Profile and Depressive Symptoms
Brief Title: Phototherapy in Young People With Depression
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Ottawa (Other)
Collaborators: University of Sydney (Other)
Responsible Party: Principal Investigator, Rébecca Robillard, Research Fellow, University of Ottawa
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015007
Record Dates: First submitted 2015-05-14; First posted 2015-05-19 (Estimated); Last update posted 2015-05-19 (Estimated); Status verified 2015-05

CONDITIONS: Depression
Keywords: Phototherapy; Light; Depression; Sleep and circadian disturbances; Youth
MeSH Terms: conditions — Depression

ARMS (1):
- Phototherapy (Other)
  Interventions: Device: Phototherapy light-emitting glasses

INTERVENTIONS:
Device: Phototherapy light-emitting glasses — The intervention consists of four weeks of bright light exposure with light-emitting glasses (blue-green 500 nm dominant wavelength; 506 Lux lm/m^2) upon awakening and progressive shift to earlier wake-up times.
  Participants are encouraged to complete the light exposure sessions for 60 min each day. Participants are also instructed to progressively shift their schedule 15 min earlier every day. This shift continues until the end of the four weeks of the intervention, or stops if the target wake-up time of 7:30am is reached (in which case, participants keep a stable wake-up and light session schedule at 7.30am for the remainder of the intervention). If participants already wake-up before 7.30am at study entry, they do the light exposure sessions upon awakening across the four weeks of the intervention.
  During the intervention, participants are asked to note down the time of each light exposure session in a diary. Adherence is also monitored and promoted through weekly phone calls.
  Other Names: Re-timer

SUMMARY:
Bright light therapy is an established treatment pathway for sleep and circadian disorders and evidence suggests that it has antidepressant effects. The underlying mechanisms of these antidepressant effects are not fully understood and results from previous studies are somewhat variable. One of the important limitations of previous depression studies has been the heterogeneity of samples in which bright light therapy has been administered.

The main aim of this study is to evaluate whether the antidepressant effects of phototherapy in young persons with depression are modulated by changes in the sleep-wake cycle. We hypothesize that more pronounce initial sleep-phase delay will predict better antidepressant response to phototherapy and that the magnitude of changes in depressive symptoms across the course of the intervention will correlate with changes in the sleep-wake cycle.

ELIGIBILITY:
Inclusion Criteria:

1. Quick Inventory of Depressive Symptomatology score > 6;
2. First episode of depression before age 25;
3. Currently engaged in, or about to start treatment for an affective disorder at a mental health clinic.

Exclusion Criteria:

1. Evidence of other sleep, neurological or primary medical conditions that could explain the current depression and/or contribute to sleep-wake dysfunction;
2. Other primary psychiatric disorders aside from anxiety disorders;
3. Significant alcohol or other substance dependence;
4. Use of medications that affect sleep, circadian rhythms, or alertness within the past month (participants stabilized on an antidepressant medication, stimulants, lithium or melatoninergic agents will not be excluded from the study);
5. Use of medications that may interact with light to produce a photoallergic reaction;
6. Eye or skin condition which may interact with bright light exposure;
7. Regular shift-work within 60-days prior to entry into the study;
8. Recent transmeridian travel.

Ages: 13 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-04; Primary Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Severity of Depression | Between baseline and post (4 weeks) intervention
  Change in severity of depression as measured by the Quick Inventory of Depressive Symptomatology (QIDSA17-SR)

SECONDARY OUTCOMES:
Severity of Depression | Score between baseline and follow up (8 weeks)
  Change in depression as measured by the Quick Inventory of Depressive Symptomatology (QIDSA17-SR)
Associations between Changes in Sleep-Wake Profile and Changes in Severity of Depression | Between baseline and post (4 weeks) intervention
  Associations between changes in sleep-wake profile (mean sleep onset time, offset time efficiency and acrophase), as measured by actigraphy, and change in depression severity as measured by the Quick Inventory of Depressive Symptomatology (QIDSA17-SR)
Associations between Initial Sleep-Wake Profile and Changes in Severity of Depression | Baseline and post (4 weeks) intervention
  Associations between the initial sleep-wake profile (mean sleep onset time, offset time efficiency and acrophase), as measured by actigraphy, and change in depression severity as measured by the Quick Inventory of Depressive Symptomatology (QIDSA17-SR)
Subjective Sleep Quality | Between baseline and post (4 weeks) intervention
  Change in Leeds Sleep Evaluation Questionnaire score
Fatigue Severity | Between baseline and post (4 weeks) intervention
  Change in Fatigue Severity Scale score

CONTACTS AND LOCATIONS:
Locations (2):
- Brain and Mind Research Insitute, The University of Sydney, Camperdown, New South Wales, Australia
- Sleep and Depression Research Units, Institute of Mental Health Research, University of Ottawa, Ottawa, Ontario, Canada